CLINICAL TRIAL: NCT04152239
Title: Prospective Evaluation of the Utility of Motorized Spiral Enteroscopy in Patients With Suspected Small Bowel Pathology
Brief Title: Utility of Motorized Spiral Enteroscopy for Suspected Small Bowel Pathology
Acronym: MSESB
Status: Terminated | Type: Observational
Why Stopped: Equipment was recalled by manufacturer and was no longer available
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Raymond Shing Yan Tang, Clinical Professional Consultant, Chinese University of Hong Kong
Other Study IDs: MSE SB study
Record Dates: First submitted 2019-11-02; First posted 2019-11-05 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Small Bowel Disease
Keywords: enteroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Study group includes consecutive patients with suspected small bowel pathology based on clinical presentation, small bowel imaging or capsule endoscopy indicated for diagnostic and/or therapeutic enteroscopy. Patients fulfilling the inclusion criteria and without exclusion criteria would undergo MSE per study protocol.
  Interventions: Procedure: Motorized spiral enteroscopy (MSE)

INTERVENTIONS:
Procedure: Motorized spiral enteroscopy (MSE) — Endoscopic Procedures MSE is a 1.6m enteroscope equipped with a single-use short spiral overtube propelled by a user-controlled motor contained in the handle of the endoscope. The endoscopist controls the left-right and up-down movements by the usual manuvers while the forward or backward advancement of the enteroscope would be contolled by a foot pedal that activates the spiral overtube rotation. Antegrade MSE, retrograde MSE, or combined antegrade and retrograde MSE would be performed as clinically indicated for diagnostic +/- therapeutic procedures.

SUMMARY:
Diagnosis and treatment of small bowel pathologies remain challenging due to the long length of the small bowel. Obscure gastrointestinal (GI) bleeding with negative upper and lower GI workup, suspected inflammatory bowel disease, and suspected tumors of the small bowel often require small bowel investigation.

While video capsule endoscopy (VCE) and computed tomography (CT) enteroclysis (CTE) are often the initial diagnostic modalities for suspected small bowel pathologies and can provide structural information of the small bowel mucosa, biopsy or therapy for the detected pathology could not be performed with VCE or CTE. In patients who require biopsy or therapy of the detected small bowel pathology, deep enteroscopy would be the procedure of choice in modern clinical practice before subjecting patient to surgery.

Diagnostic and therapeutic deep enteroscopy can be performed by balloon overtube assisted enteroscopy (eg, double balloon enteroscopy (DBE), single balloon enteroscopy (SBE) or spiral overtube assisted enteroscopy (SE). Despite the difference in equipment design of DBE, SBE, and SE, the concepts for small bowel intubation by pleating the intestine over the endoscope are the same behind these techniques. Depending on the location of the small bowel pathology reported by VCE or CTE, antegrade (oral route), retrograde (anal route), or combined antegrade and retrograde deep enteroscopy for total enteroscopy can be performed.

DETAILED DESCRIPTION:
Diagnosis and treatment of small bowel pathologies remain challenging due to the long length of the small bowel. Obscure gastrointestinal (GI) bleeding with negative upper and lower GI workup, suspected inflammatory bowel disease, and suspected tumors of the small bowel often require investigations of the small bowel.

While video capsule endoscopy (VCE) and computed tomography (CT) enteroclysis (CTE) are often the initial diagnostic modalities for suspected small bowel pathologies and can provide structural information of the small bowel mucosa, biopsy or therapy for the detected pathology could not be performed with VCE or CTE. In patients who require biopsy or therapy of the detected small bowel pathology between the ligament of Treitz and ileocecal valve, deep enteroscopy would be the procedure of choice in modern clinical practice before subjecting patient to surgery.

Diagnostic and therapeutic deep enteroscopy can be performed by balloon overtube assisted enteroscopy (eg, double balloon enteroscopy (DBE), single balloon enteroscopy (SBE) or spiral overtube assisted enteroscopy (SE)). Despite the difference in equipment design of DBE, SBE, and SE, the concept for small bowel intubation by pleating the intestine over the endoscope is the same behind these techniques. Depending on the location of the small bowel pathology reported by VCE or CTE, antegrade (oral route), retrograde (anal route), or combined antegrade and retrograde deep enteroscopy for total enteroscopy can be performed. In patients with suitable anatomy, total enteroscopy by antegrade approach alone may be achieved.

DBE was introduced in 2001 and has been the most studied form of modern deep enteroscopy. In a recent systematic review of 12823 procedures, the overall diagnostic yield was found to be 68.1%. The pooled total enteroscopy rate was 44% by the combined anterograde and retrograde approach or antegrade-only approach. The pooled minor and major adverse event (eg, perforation, bleeding, pancreatitis, aspiration pneumonia) rates were 9.1% and 0.72%, respectively. Despite its clinical utility, long procedure time (usually more than 1 to 1.5 hour) and the need for 2-operators are often regarded as drawbacks of DBE. SE was subsequently designed to address this issue with the use of a spiral overtube by manual rotation for efficient small bowel intubation. When compared to balloon overtube assisted enteroscopy, the main advantage of SE is the relative reduction in procedure time. However, the total enteroscopy rate of SE is lower, mainly due to difficult overtube and endoscope passage in retrograde procedures. Adverse events with SE (eg, minor mucosal tears, perforation, etc) have been reported to be 0.3%. Because both DBE and SE have its own shortcomings, the need to further improve the current technology of deep enteroscopy has always been present.

Recently, a motorized spiral enteroscope (MSE) (Olympus Medical, Tokyo, Japan) has become available and has the potential to address the shortcomings of the DBE and SE. MSE is an enteroscope equipped with a short spiral overtube propelled by a endoscopist-controlled motor contained in the handle of the endoscope. The endoscopist controls the left-right and up-down movements by the usual manuvers while the forward or backward advancement of the enteroscope would be contolled by a foot pedal that activates the spiral overtube rotation. The basic principle of small bowel pleating over the endoscope by the use of an overtube to achieve deep small bowel intubation is similar to that of DBE and SE. During the procedure, a visual force gauge allows the operator to monitor the direction of overtube rotation and the resistance applied to the spiral overtube in the small bowel. If excessive rotational resistance is detected, the motor would be stopped automatically to avoid mucosal trauma in the intestine. The initial experience of MSE in patients with small bowel pathology and colonic pathology appears promising with a diagnostic yield of 76 - 88%, therapeutic yield of 76%, a total enteroscopy rate of 70% (combined antegrade and retrograde approaches or antegrade alone approach) and shorter procedure time (< 40 minutes). Based on data from three studies including a total of 110 MSE procedures, no serious adverse event such as perforation has been reported. The overall adverse event rate including erosion, mucosal tear, hematoma, transient swallowing discomfort, etc, was reported to be 20% in a study with 30 patients. Despite its potential to improve the clinical management of patients with small bowel disorders, current data on the diagnostic and therapeutic utility of MSE is from expert European centers and remains limited. Investigators therefore propose this study to evaluate the utility of the MSE in patients with suspected small bowel pathology.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients with suspected small bowel pathology based on clinical presentation, small bowel imaging or capsule endoscopy indicated for diagnostic and/or therapeutic enteroscopy
* Written informed consent available

Exclusion Criteria:

* Contraindications for endoscopy due to comorbidities
* Unable to provide written informed consent
* Patients with known severe GI tract inflammation, intestinal obstruction, gastroesophageal varices that preclude a safe enteroscopy procedure
* Coagulopathy or thrombocytopenia that cannot be corrected by blood product transfusion
* Pregnant patients
* Moribund patients from terminal illnesses

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with suspected small bowel pathology indicated for deep enteroscopy for diagnostic +/- therapeutic procedure.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield | peri-procedure
  Diagnostic yield: defined as successful identification of the suspected pathology based on clinical presentation, pre-MSE small bowel imaging or capsule endoscopy

SECONDARY OUTCOMES:
Technical success | peri-procedure
  - defined as successful advancement of enteroscope beyond the ligament of Treitz for antegrade procedures, or successful advancement of enteroscope proximal to the ileocecal valve for retrograde procedures
Therapeutic yield | peri-procedure
  Therapeutic yield: defined as successful endoscopic interventions such as treatment for GI bleeding, polypectomy, etc
Insertion time | peri-procedure
  Insertion time: defined as time to the maximal depth of insertion in small bowel
Maximal depth of insertion in small bowel | peri-procedure
  Maximal depth of insertion in small bowel
Rate of total enteroscopy | peri-procedure
  Rate of total enteroscopy achieved by antegrade approach alone or combined antegrade and retrograde approaches if total enteroscopy is indicated by findings on pre-MSE small bowel imaging or capsule endoscopy
Adverse events related to procedure | peri-procedure
  Adverse events related to procedure

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Tang, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, The Chinese University of Hong Kong, Shatin, New Territories, Hong Kong